CLINICAL TRIAL: NCT00253240
Title: Diabetes Screening, Risk Management and Disease Management in a High-Risk Mental Health Population - An Evaluation Project
Brief Title: Diabetes Screening, Risk Management and Disease Management in a High-Risk Mental Health Population
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government); Western Ontario Therapeutic Community Hostel (WOTCH) (Unknown); Canadian Mental Health Association (Other); London Intercommunity Health Centre (LIHC) (Other)
Responsible Party: Sponsor
Other Study IDs: R-04-441; G13-05457; 10933E; LRI7760576
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Diabetes Mellitus; Schizophrenia; Psychotic Disorders
MeSH Terms: conditions — Diabetes Mellitus; Schizophrenia; Psychotic Disorders | interventions — Mass Screening; Therapeutics

STUDY DESIGN:
Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Screening
Procedure: Management

SUMMARY:
Family physicians are the primary health care providers for complex patients such as persons with serious mental illness. The psychiatric needs of these patients could take attention away from management of health problems and from usual health promotion services. For example, Schizophrenia is associated with a higher than normal incidence of diabetes, and first line treatments of Schizophrenia have also been found to increase risk for diabetes. As such, this high-risk group requires targeted diabetes strategies. In London Ontario, services are provided to this high risk mental health population primarily by two community agencies: The Western Ontario Therapeutic Community Hostel (WOTCH) and the Canadian Mental Health Association (CMHA). Accordingly, the goal of this project is to assess how these patients are currently being managed by their family physicians and to pilot a community-based, multidisciplinary diabetes clinic model within this population. If this delivery model proves feasible and effective, family physicians could be assisted by existing community agencies in the management of their patients' diabetes and patients will receive improved access to this vital multidisciplinary team.

DETAILED DESCRIPTION:
In London Ontario, community based services are provided to the high-risk mental health population by primarily two community agencies: The Western Ontario Therapeutic Community Hostel (WOTCH) and the Canadian Mental Health Association (CMHA). WOTCH provides treatment, support, rehabilitation and recovery services to individuals with serious mental illness including case management, social recreational activities, and vocational and housing options. Each client is linked to a Community Support Worker who meets with the clients in their homes or in other community locations to develop rehabilitation plans, monitor the success of these plans, coordinate services and advocate on the client's behalf. Similarly, CMHA provides a range of education and support services in the London Middlesex area. CMHA provides centralized Intake and Assessment for WOTCH, London East Community Mental Health Services and for their own Community Support Case Management program. The qualifying criteria for access to the programs are based on assessment of three key elements: Disability, Duration and Dysfunction.

Collectively WOTCH, CMHA and the London Mental Health Crisis Service maintain a common client record for clients. Individuals generate crisis plans and information is attained which includes primary diagnosis, co-morbid health conditions, medication, demographics and family physician.

Project Population -

Participants in the project were drawn from the active WOTCH and CMHA database. Participants that were identified in the database as having a diagnosis of Schizophrenia (or Psychotic Disorder) and/or treatment with a Novel Antipsychotic medication were approached for participation in the project. Any participants identified in the database with a pre-existing diagnosis of diabetes were not included in the initial selection of participants. A total of 60 participants meeting the above criteria were selected for the initial screening phase of the project.

Phase One

The first phase of the proposed project aims to determine how these complex patients were being managed in primary care. Consent was sought from family physicians that were determined to be the primary care providers for the participants who met criteria for involvement in the project. A chart review was conducted on site at each family practice location in a space provided by the physician. The review includes demographic information, diagnoses, medication use (past and current), lab results (blood glucose and lipid profile), and a medication side effects profile.

Phase Two

The second phase of the proposed project aims to quantify the prevalence and risk profile of diabetes mellitus, as well as mental illness symptomology and disability, in this identified high-risk population. All participants identified in the chart review as not having received an Oral Glucose Tolerance Test (OGTT) in the past year, in accordance with current guidelines, were followed in phase two of the proposed project. In addition, caseworker feedback was used as a source of information regarding prior screening in cases where physicians did not consent to participate in the chart audit but the client did consent to participate. Participants identified as being in need of an OGTT for screening of DM were invited to attend a screening event held at CMHA or WOTCH facilities. Caseworkers played an active role in facilitating participants' attendance at the screening events. A phlebotomy certified staff member conducted the OGTT's. If a lipid profile had not been completed within the past year, the current sample will also be analyzed for lipids. Diabetes risk profile, the Brief Symptom Inventory (BSI) and the World Health Organization Disability Scale (WHO-DAS II) were also completed at this time. The OGTT was sent by the phlebotomist to a major central lab, contracted by the project, to ensure internal consistency of the analyses. Copies of the lab results were sent to the family physician, for placement in the participants' file, and to the data manager, for analyses related to the proposed study.

Phase Three

The third phase of the proposed project aims to evaluate the implementation of a multidisciplinary model of care, consistent with current guidelines for diabetes management, within this high-risk population. Participants identified in either of the previous two phases as having diabetes or pre-diabetes were invited to participate in a multidisciplinary program for diabetes management. The program runs monthly at identified usual point of WOTCH and CMHA service locations. Identified WOTCH and CMHA staff are encouraged to attend the program to serve as a consistent source of progress monitoring and to increase their knowledge and familiarity with the goals of diabetes management and diabetes complications. The program is based on the London Intercommunity Health Centre's (LIHC) diabetes risk and disease management program previously piloted within a Community Health Centre. During the clinic, participants meet individually with the Nurse Practitioner (NP) who works through a Diabetes Care Flow Sheet. At each monthly visit, the NP assesses glycemic control, hypertension, medications, weight, and foot care. Lifestyle counseling is also provided with respect to smoking, activity, diet and stress. At each participant's initial visit, he or she is provided with a pedometer and instructed on its use. This aids the NP in assessing physical activity and provides a motivational tool for the participant. The NP is responsible for highlighting any variables that fall outside the expected range. If it is decided that there are issues that need further clinical consultation, the NP then refers the participant to the appropriate team member. The DHC team includes a foot care specialist, dietician, Diabetes Education Nurse, and a family physician. The family physician team leader refers any clinical issues that fall beyond the scope of the DHC for specialist follow up. Each participant receives appropriate instructions regarding return to the multidisciplinary clinic.

The NP also monitors each participant's need for periodic lab testing of glucose and lipids. Annual screening for neuropathy, nephropathy, and eye exams are indicated on the Diabetes Care Flow Sheet. The DHC team sends participants' family physicians' reminder notices of these regularly needed referrals as well as any relevant clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Active in current WOTCH/CMHA database with listed diagnosis of a psychotic disorder an or use of Novel Antipsychotics. Must have Family Physician contact.

Exclusion Criteria:

* any patient with declaration on file stating incapable of consenting to treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2004-09 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David RS Haslam, MSc MD FRCPC, Principal Investigator — St. Joseph's Health Care London; Stewart B Harris, MD MPH CCFP FACPM, Principal Investigator — Centre for Studies in Family Medicine
Locations (1):
- London Intercommunity Health Centre, London, Ontario, Canada